CLINICAL TRIAL: NCT03011736
Title: Single-Arm, Non-inferiority Study of Omission of Intraoperative Intact Parathyroid Hormone (PTH) During Minimally Invasive Parathyroidectomy for Primary Hyperparathyroidism
Brief Title: Omission of Intact Parathyroid Hormone Testing During Surgery in Treating Patients With Primary Hyperparathyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 274915; NCI-2016-01974 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 274915 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Parathyroid Gland Adenoma; Primary Hyperparathyroidism
MeSH Terms: conditions — Parathyroid Neoplasms; Hyperparathyroidism, Primary | interventions — Parathyroidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive Care (parathyroidectomy) (Experimental): Patients undergo standard minimally invasive parathyroidectomy without PTH testing during surgery.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Parathyroidectomy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Parathyroidectomy — Undergo parathyroidectomy

SUMMARY:
This clinical trial studies the omission of intact parathyroid hormone testing during surgery in treating patients with primary hyperparathyroidism. Omission of intact parathyroid hormone testing during parathyroid gland removal may help patients with primary hyperparathyroidism to decrease their time under anesthesia, and decrease the overall time and cost of surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the non-inferiority of omission of parathyroid hormone (PTH) in patients who meet the biochemical and radiological criteria compared to current standard of care (i.e. use of intraoperative parathyroid hormone testing).

SECONDARY OBJECTIVES:

I. Cost-analysis to determine savings of omission of intraoperative PTH testing.

OUTLINE:

Patients undergo standard minimally invasive parathyroidectomy without PTH testing during surgery.

After completion of study, patients are followed up at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Positive 4 dimensional computed tomography (4D CT) for single gland (adenoma) primary hyperparathyroidism
* Preoperative serum calcium levels >= 10.9 mg/dL
* Preoperative parathyroid hormone (PTH) elevated beyond normal range or inappropriately high for associated calcium level
* Patient has no history of prior neck surgery or external radiation to neck for malignant conditions
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patient has recurrent hyperparathyroidism
* 4D CT positive for multiple gland disease
* Patient has inability to tolerate 4D CT scan (for example; contrast intravenous (IV) allergy, claustrophobia, renal disease)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female subjects; may be determined in the preoperative evaluation
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the subject an unsuitable candidate to undergo observational study (may also include preoperative testing results including electrocardiography [EKG], chest x-ray, or pulmonary function tests that preclude a wide excision in the operating room)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Cure of primary hyperparathyroidism following surgery with intraoperative PTH omission | At 2 weeks
  Will be evaluated using a binomial exact test. If all N=60 patients achieve cure then the proposed surgery with intraoperative PTH testing committed will be considered non inferior. A 95% confidence interval about pi will be obtained.

SECONDARY OUTCOMES:
Post-operative cost analysis | At 2 weeks
  cost analysis will be based on operative time and omission of intraoperative PTH levels.

CONTACTS AND LOCATIONS:
Overall Officials: Moshim Kukar, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States